CLINICAL TRIAL: NCT00615004
Title: An Observational, Retrospective, Comparative Study to Investigate Differential Outcome on Cardiomyopathy Following Control of Acromegaly After Surgery or Somatostatin Analogues Given as First-Line Therapy
Brief Title: Cardiovascular Outcome After Surgery or Somatostatin Analogues
Acronym: CVAcro
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Annamaria Colao, Department of Molecular and Clinical Endocrinology and Oncology
Other Study IDs: NeuroendoUnit-7
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2008-02-14 (Estimated); Status verified 2007-12

CONDITIONS: Acromegaly
Keywords: Acromegaly; GH; IGF-I; Octreotide-LAR; Lanreotide; Transsphenoidal surgery
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Sera from most patients on a yearly bases are stored in our freezed at minus 80° for eventual further studies. No experimental parameters are included in the current study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1-SSA: All patients receiving first-line depot SSA treatment, with either octreotide-LAR or lanreotide, achieving control of the disease, and with available follow-up after 12 months of treatment.
- 2-Surgery: All patients treated with first-line surgery via trans-sphenoidal route by microscopic and/or endoscopic approach, who did not require any additional therapy for acromegaly and with available follow-up after 12 months of treatment

SUMMARY:
A direct comparison between the results of surgery or somatostatin analogues (SSA) on cardiovascular complication in acromegaly has never been performed.

Our objective is to investigate whether first-line surgery or SSA have a different outcome on cardiomyopathy after 12 months. The design of the study is retrospective, comparative, non randomized, because of ethical problems.

Setting University Hospital. All patients treated with SSA [either octreotide-LAR (10-40 mg/q28d), or lanreotide (30-120 mg/q28d); dosages up-titrated to control GH and IGF-I levels] or operated on by transsphenoidal approach. For the purposes of this study only controlled patients will be included.

Measurements Primary outcome measures were changes in left ventricular mass index (LVMi), diastolic [early to atrial mitral flow velocity (E/A)] and systolic perform-ance [LV ejection fraction (LVEF)]. Secondary outcome measures were reduction of total/HDL-cholesterol ratio, as a cardiovascular (CV) risk parameter, improvement of glucose profile and pituitary function, as indirect causes of CV improvement.

Expected results: SSA and surgery groups should have similar results in terms of improvement of cardiomyopathy. However, recent data suggest that SSA reduce directly heart rate and cardiomyocytes performance: clinical implications of these evidences suggest that SSA will improve cardiovascular outcome more than surgery. Moreover, after surgery, replacement therapy already stabilised or of new onset, has never been considered so far in this setting.

DETAILED DESCRIPTION:
We will review all files from consecutive patients with active acromegaly coming to the Units of Endocrinology or Neurosurgery of the "Federico II" University of Naples from Jan 1st 1997 to December 31st 2006, primarily treated with either surgery or depot SSA, i.e. lanreotide (LAN) or slow-release octreotide (LAR), and with an available follow-up of at least 12 months. Due to the study design, this is a non randomized study. However, our routine procedure generally considers first-line treatment with SSA for 6-12 months, unless the tumors are clearly non invasive on Magnetic Resonance Imaging (MRI) and/or the patients who do not present any surgical or anesthesiological risk.

Cure criteria are considered according with Giustina et al. Acromegaly is considered to be controlled if mean fasting GH levels were ≤2.5 μg/liter in presence of normal IGF-I levels for sex and age. Nadir GH after oral glucose load (oGTT) ≤1 μg/liter is also an option to evaluate disease control according with the 2000 Consensus Statement. However, oGTT is generally not routinely performed in patients receiving SSA, since GH-induced glucose suppression is likely to be mediated by the endogenous somatostatin tone. To avoid ascertainment bias, disease control after surgery and SSA will be only based on fasting GH and IGF-I levels. The diagnosis of acromegaly is defined as previously reported, by high serum GH levels during a 6 hr time course, not suppressible <1 µg/l after oGTT and high plasma IGF-I levels for age [expressed as value upper limit of normal range (ULN)].

For the purpose of this study only the patients with controlled acromegaly will be included to provide a period of follow-up long enough to investigate changes in cardiomyopathy parameters.

Study protocol: As for our routine procedure, at diagnosis all the patients undergo a complete metabolic and endocrine screening. After an overnight fasting, serum IGF-I levels are assayed twice in a single sample at the time 0 of the GH profile; GH levels are calculated as the mean value of at least 5 (up to 8) samples drawn every 30 min over a period of three-six hours and the average value will be considered for the statistical analysis; fasting total cholesterol, HDL cholesterol, glucose and insulin levels are also measured. The total/HDL-cholesterol ratio, index of cardiovascular risk, is calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with first-line surgery via trans-sphenoidal route by microscopic and/or endoscopic approach or with first-line depot SSA treatment
* Achieving control of the disease; AND
* With available follow-up after 12 months of treatment

Exclusion Criteria:

* Patients receiving second surgery within 3 months from first surgery
* Requiring combined dopamine-agonists and SSA because of a mixed GH/PRL-secreting tumor
* Receiving the s.c. octreotide for longer than 15 days; OR
* Requiring surgery or SSA as second-line treatment before the completion of the 12 months or with a follow-up shorter than 6 months after surgery or pharmacotherapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will review all files from consecutive patients with active acromegaly coming to the Units of Endocrinology or Neurosurgery of the "Federico II" University of Naples from Jan 1st 1997 to December 31st 2006, primarily treated with either surgery or depot SSA, i.e. lanreotide (LAN) or slow-release octreotide (LAR), and with an available follow-up of at least 12 months. Due to the study design, this is a non ran-domized study. However, our routine procedure generally considers first-line treatment with SSA for 6-12 months, unless the tumors are clearly non invasive on Magnetic Resonance Imaging (MRI) and/or the patients who do not present any surgical or anesthesiological risk.
Sampling Method: Probability Sample
Enrollment: 215 (Actual)
Dates: Start 1997-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Changes of left ventricular mass index (LVMi), as measure of LV hypertrophy, early to atrial mitral flow velocity (E/A), as measure of diastolic function, and left ventricular ejection fraction (LVEF), as measure of systolic function. | 12 months

SECONDARY OUTCOMES:
Changes in the total/HDL cholesterol ratio, glucose tolerance, measured as fasting glucose levels and HOMA reduction, and improvement of pituitary function | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Colao, MD, Principal Investigator — Federico II University
Locations (1):
- Department of Molecular and Clinical Endocrinology and Oncology, University Federico II of Naples, Naples, Naples, Italy

REFERENCES:
- [Result] Colao A, Lombardi G. Growth-hormone and prolactin excess. Lancet. 1998 Oct 31;352(9138):1455-61. doi: 10.1016/S0140-6736(98)03356-X. PMID 9808008
- [Result] Melmed S. Medical progress: Acromegaly. N Engl J Med. 2006 Dec 14;355(24):2558-73. doi: 10.1056/NEJMra062453. No abstract available. PMID 17167139
- [Result] Melmed S, Casanueva F, Cavagnini F, Chanson P, Frohman LA, Gaillard R, Ghigo E, Ho K, Jaquet P, Kleinberg D, Lamberts S, Laws E, Lombardi G, Sheppard MC, Thorner M, Vance ML, Wass JA, Giustina A. Consensus statement: medical management of acromegaly. Eur J Endocrinol. 2005 Dec;153(6):737-40. doi: 10.1530/eje.1.02036. PMID 16322377
- [Result] Sheppard MC. Primary medical therapy for acromegaly. Clin Endocrinol (Oxf). 2003 Apr;58(4):387-99. doi: 10.1046/j.1365-2265.2003.01734.x. PMID 12641619
- [Result] Giustina A, Barkan A, Casanueva FF, Cavagnini F, Frohman L, Ho K, Veldhuis J, Wass J, Von Werder K, Melmed S. Criteria for cure of acromegaly: a consensus statement. J Clin Endocrinol Metab. 2000 Feb;85(2):526-9. doi: 10.1210/jcem.85.2.6363. PMID 10690849
- [Result] Colao A, Martino E, Cappabianca P, Cozzi R, Scanarini M, Ghigo E; A.L.I.C.E. Study Group. First-line therapy of acromegaly: a statement of the A.L.I.C.E. (Acromegaly primary medical treatment Learning and Improvement with Continuous Medical Education) Study Group. J Endocrinol Invest. 2006 Dec;29(11):1017-20. doi: 10.1007/BF03349217. No abstract available. PMID 17259801
- [Result] Cappabianca P, Alfieri A, Colao A, Ferone D, Lombardi G, de Divitiis E. Endoscopic endonasal transsphenoidal approach: an additional reason in support of surgery in the management of pituitary lesions. Skull Base Surg. 1999;9(2):109-17. doi: 10.1055/s-2008-1058157. PMID 17171126
- [Result] Galderisi M, Vitale G, Bianco A, Pivonello R, Lombardi G, Divitiis Od, Colao A. Pulsed tissue Doppler identifies subclinical myocardial biventricular dysfunction in active acromegaly. Clin Endocrinol (Oxf). 2006 Apr;64(4):390-7. doi: 10.1111/j.1365-2265.2006.02475.x. PMID 16584510
- [Result] Colao A, Pivonello R, Rosato F, Tita P, De Menis E, Barreca A, Ferrara R, Mainini F, Arosio M, Lombardi G. First-line octreotide-LAR therapy induces tumour shrinkage and controls hormone excess in patients with acromegaly: results from an open, prospective, multicentre trial. Clin Endocrinol (Oxf). 2006 Mar;64(3):342-51. doi: 10.1111/j.1365-2265.2006.02467.x. PMID 16487447
- [Result] Colao A, Ferone D, Marzullo P, Lombardi G. Systemic complications of acromegaly: epidemiology, pathogenesis, and management. Endocr Rev. 2004 Feb;25(1):102-52. doi: 10.1210/er.2002-0022. PMID 14769829
- [Derived] Colao A, Auriemma RS, Savastano S, Galdiero M, Grasso LF, Lombardi G, Pivonello R. Glucose tolerance and somatostatin analog treatment in acromegaly: a 12-month study. J Clin Endocrinol Metab. 2009 Aug;94(8):2907-14. doi: 10.1210/jc.2008-2627. Epub 2009 Jun 2. PMID 19491229
- [Derived] Colao A, Pivonello R, Galderisi M, Cappabianca P, Auriemma RS, Galdiero M, Cavallo LM, Esposito F, Lombardi G. Impact of treating acromegaly first with surgery or somatostatin analogs on cardiomyopathy. J Clin Endocrinol Metab. 2008 Jul;93(7):2639-46. doi: 10.1210/jc.2008-0299. Epub 2008 Apr 29. PMID 18445662